CLINICAL TRIAL: NCT02952677
Title: "Remind-to-move" Using Wearable Devices in Home-based Treatment for Promoting Upper Extremity Recovery in Patients With Stroke After Subacute Discharge
Brief Title: "Remind-to-move" for Promoting Upper Extremity Recovery in Patients With Stroke After Subacute Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Tuen Mun Hospital (Other Government); Kowloon Hospital, Hong Kong (Other); Guangzhou First People's Hospital (Other); Guangzhou Panyu Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRF/5608/12M
Record Dates: First submitted 2016-08-31; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-08

CONDITIONS: Stroke; Upper Extremity Hemiplegia
MeSH Terms: conditions — Stroke | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental (Experimental): Participants receive "Remind-to-move" by means of vibration emitted through sensory cueing wristwatch devices, 3 consecutive hours daily, for 4 weeks, as well as usual care during the intervention period.They are also encouraged to use their arms as much as possible and the accelerometer built-in the device record the arm movement during daily activities.
  Interventions: Behavioral: Remind-to-move; Other: Control
- Sham treatment (Sham Comparator): Participants wear sham wristwatch devices but without vibration cueing, 3 consecutive hours daily, for 4 weeks, as well as usual care during the intervention period. They are also encouraged to use their arms as much as possible and the accelerometer built-in the device record the arm movement during daily activities.
  Interventions: Behavioral: Sham; Other: Control
- Control (Other): Participants receive usual care only during the intervention period.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Remind-to-move — Participants were required to wear sensory cueing wristwatch devices with vibration emitted on the affected arm for 3 consecutive hours daily, for a total of 4 weeks, at any time during the day, and received usual care as well.
  Other Names: Sensory cueing
  Arms: Experimental
Behavioral: Sham — Participants were required to wear sensory cueing wristwatch devices without vibration emitted on the affected arm for 3 consecutive hours daily, for a total of 4 weeks, at any time during the day, and received usual care as well.
  Arms: Sham treatment
Other: Control — Participants received usual care

SUMMARY:
This is a multi-centered randomized controlled trial to investigate the effects of "Remind-to-Move" (RTM) using wearable devices at home for promoting upper extremity recovery in stroke patients after discharge from subacute hospitals.

DETAILED DESCRIPTION:
This is a proof-of-principle study to investigate the effects of "Remind-to-Move" (RTM) using wearable devices at home for promoting upper extremity recovery in stroke patients after discharge from subacute hospitals.

A multi-center, parallel-group, randomized controlled trial with blinded assessment was carried out in four hospitals. Eighty-four eligible participants who had suffered from stroke with less than 6 months and could slightly move their arms were randomly allocated to either an experimental, sham, or control group stratified by hemiplegic arm functional levels. Patients in the experimental group were treated by RTM using wearable devices, 3 consecutive hours daily, for 4 weeks. The sham group used sham devices. The control group received the usual care. A masked assessor evaluated the participants at 0, 4th, 8th and 12th weeks. Outcome measures included arm function tests, motor activity log, movement amount and percentage recorded by wearable devices. All patients allocated to treatment were included in intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Frst-time ischemic or hemorrhagic stroke confirmed by magnetic resonance imaging or X-ray computed tomography
2. Unilateral hemispherical involvement
3. Aged 18 or above
4. Time since onset less than 6 months
5. Functional Test for Hemiplegic Upper Extremity Hong Kong version (FTHUE-HK) ≥ 3 (maximum 7)
6. Able to understand verbal instruction and follow one-step commands
7. Modified Ashworth Scale (MAS) ≤ 2
8. Mini-mental State Examination (MMSE) ≥ 19
9. No complaint of excessive pain or swelling over hemiplegic arm
10. Sensation on the affected wrist intact or with mild impairment only (National Institute of Health Stroke Scale=0 or 1).

Exclusion Criteria:

1. Participating in any experimental or drug study
2. Unable to give consent to participate
3. Of inadequate balance as indicated by the inability to stand for at least 2 minutes with or without arm support
4. Having history of botulinum toxin injection in 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-11; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment-Upper Extremity Score | Change from Baseline to 4-week, plus follow-ups at 8-week and 12-week
  Hemiplegic arm motor impairment scale

SECONDARY OUTCOMES:
Functional Independence Measure | Change from Baseline to 4-week, plus follow-ups at 8-week and 12-week
  Self-care performance scale
Motor Activity Log | Change from 4-week to follow-ups at 8-week and 12-week
  Daily activity log
Accelerometry in wristwatch devices | Change from Baseline to 4-week
  Kinematic data recorded by the built-in accelerometers
Box and Block Test | Change from Baseline to 4-week, plus follow-ups at 8-week and 12-week
  Hemiplegic arm laboratory dexterity test
Action Research Arm Test | Change from Baseline to 4-week, and follow-ups at 8-week and 12-week
  Hemiplegic arm laboratory functional test

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth NK Fong, PhD, Principal Investigator — The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fong KN, Lo PC, Yu YS, Cheuk CK, Tsang TH, Po AS, Chan CC. Effects of sensory cueing on voluntary arm use for patients with chronic stroke: a preliminary study. Arch Phys Med Rehabil. 2011 Jan;92(1):15-23. doi: 10.1016/j.apmr.2010.09.014. PMID 21187201
- [Background] Fong KN, Yang NY, Chan MK, Chan DY, Lau AF, Chan DY, Cheung JT, Cheung HK, Chung RC, Chan CC. Combined effects of sensory cueing and limb activation on unilateral neglect in subacute left hemiplegic stroke patients: a randomized controlled pilot study. Clin Rehabil. 2013 Jul;27(7):628-37. doi: 10.1177/0269215512471959. Epub 2013 Feb 12. PMID 23405025